CLINICAL TRIAL: NCT06084962
Title: A Study of DeepTag-GPRC5D Targeted CAR-T Cells Therapy for Refractory/Relapsed Multiple Myeloma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: He Huang (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Sponsor-Investigator, He Huang, Clinical Professor, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TXB2023018
Record Dates: First submitted 2023-10-10; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-09

CONDITIONS: Relapse/Refractory Multiple Myeloma
Keywords: Multiple Myeloma; DeepTag-GPRC5D CAR T-cell
MeSH Terms: conditions — Recurrence; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Administration of DeepTag-GPRC5D Targeted CAR T-cells (Experimental): Dose escalation follows the standard 3+3 dose escalation design. A total of 3 dose levels are set for subjects.
  Interventions: Biological: DeepTag-GPRC5D Targeted CAR T-cells

INTERVENTIONS:
Biological: DeepTag-GPRC5D Targeted CAR T-cells — Each subject receive DeepTag-GPRC5DTargeted CAR T-cells by intravenous infusion
  Other Names: DeepTag-GPRC5D Targeted CAR T-cells injection

SUMMARY:
Clinical Trial for the safety and efficacy of DeepTag-GPRC5D targeted CAR-T cells therapy for refractory/relapsed multiple myeloma

DETAILED DESCRIPTION:
In this study, 60 patients with relapsed refractory multiple myeloma were proposed to undergo DeepTag-GPRC5D CAR-T cell therapy. Under the premise that its safety has been clarified in previous studies, further observation and evaluation of the effectiveness of DeepTag-GPRC5D CAR-T cell therapy for relapsed refractory multiple myeloma; At the same time, on the basis of expanding the sample size, more safety data on DeepTag-GPRC5D CAR-T cell treatment for relapsed refractory multiple myeloma were accumulated, including rare and delayed complications.

ELIGIBILITY:
Inclusion Criteria:

* 1. Those who voluntarily participated in this trial and provided informed consent;
* 2. Gender unlimited，18<Age≤75;
* 3. Estimated life expectancy of minimum of 12 weeks;
* 4. ECOG 0-2;
* 5. Diagnosed as multiple myeloma according to the IMWG criteria;
* 6. Subjects failed treatment with at least 3 prior lines of therapy (including chemotherapy based on proteasome inhibitors (PIs) ，immunomodulatory agents (IMiDs) and CD38 antibody）, or recived the above three treatment methods experienced disease progression or recurrence during the most recent treatment process or within 6 months after the end of treatment, Difficulty in treatment includes primary difficulty in treatment ( patient has not achieved minimal remission or disease progression during treatment) or secondary difficulty in treatment (patient develops disease progression within 60 days after completion of treatment);
* 7. Women have a negative urine pregnancy test before the start of medication administration and agree to take effective contraceptive measures during the trial period until the last follow-up;
* 8. The blood routine meets the following standards:

  1. Lymphocyte count>0.3×10e9/L;
  2. Neutrophils ≥0.5×10e9/L;
  3. Hemoglobin ≥60g/L;
  4. Platelet ≥30×10e9/L

Exclusion Criteria:

* 1. History of craniocerebral trauma, conscious disturbance, epilepsy, cerebrovascular ischemia, and cerebrovascular hemorrhagic diseases;
* 2. Electrocardiogram shows prolonged QT interval, severe heart diseases such as severe arrhythmia in the past;
* 3. Pregnant (or lactating) women;
* 4. Patients with HIV infection;
* 5. Active infection of hepatitis B virus or hepatitis C virus;
* 6. Concurrent therapy with systemic steroids within 2 weeks prior to screening, except for the patients recently or currently receiving in haled steroids;
* 7. The proiferation rate is less than 5 times response to CD3/CD28 co-stimulation signal;
* 8. Creatinine>2.5mg/dl, or ALT / AST > 3 times of normal amounts, or bilirubin>2.0 mg/dl;
* 9. Any situations that the investigator believes may increase the risk of patients or interfere with the results of study;
* 10. Patients who received anti-cancer chemotherapy or other medications within 2 weeks before screening;
* 11. Uncontrolled malignant tumors except MM, excluding malignant tumors that received radical treatment and no active disease was found within 3 years before enrollment;
* 12. Patients who received autologous hematopoietic stem cell transplantation (ASCT) within 8 weeks before screening, or who plan to undergo ASCT during the study period;
* 13. Patients received allogeneic stem cell therapy;
* 14. Any unsuitable to participate in this trial judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-20 (Estimated); Primary Completion 2026-10-20 (Estimated); Study Completion 2026-10-20 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Up to 28 years after Treatment
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Incidence of treatment-emergent adverse events (TEAEs) | Up to 2 years after Treatment
  Incidence of treatment-emergent adverse events [Safety and Tolerability]

SECONDARY OUTCOMES:
Multiple Myeloma (MM), Overall response rate (ORR) | Up to 2 years after Treatment
  Assessment of ORR (ORR = sCR+CR+VGPR+PR+MR)
Progression-free survival (PFS) | Up to 2 years after Treatment
  The time from randomization or start of study treatment until objective tumor progression or death
Duration of remission,DOR | Up to 1 years after Treatment
  The time from CR/CRi and PR to disease relapsed or death due to disease

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, MD, Principal Investigator — Zhejiang University
Locations (1):
- The first affiliated hospital of medical college of zhejiang university, Hangzhou, Zhejiang, China